CLINICAL TRIAL: NCT04333940
Title: Impact of Periapical Radiography and Cone Beam Computed Tomography on Periapical Assessment Following Surgical Endodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dr. G.Keerthana
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Periapical Diseases
MeSH Terms: conditions — Periapical Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. 3D CBCT GROUP (Experimental): Preoperative 3-dimensional CBCT will be taken.
  Interventions: Procedure: periapical surgery
- 2D PR GROUP (Active Comparator): Preoperative 2-dimensional periapical radiographs will be taken using paralleling technique with customized Jig
  Interventions: Procedure: periapical surgery

INTERVENTIONS:
Procedure: periapical surgery — clinical signs and symptoms, probing depth, Clinical attachment level (CAL ), dimensions of lesion, distance from the defect and apex of tooth to the anatomical structures will be measured

SUMMARY:
This study will compare Cone beam Computed Tomography and Periapical radiography in detection and measurement of periapical lesions and healing outcomes following periapical surgery.

DETAILED DESCRIPTION:
Study will be conducted in Post Graduate Institute of Dental Sciences, Rohtak in the department of Conservative Dentistry & Endodontics.

Study Design: - Prospective clinical trial

Time Frame: - Jan 2019 to April 2020

Population / Participants: -Patients of age 18 years and above will be enrolled in the study.

Sample size: - The anticipated change in treatment plan was expected to be 53% before and after using CBCT. Based on the available data , sample size was calculated to enroll a minimum of 18 patients in each group with a power level of 90% and alpha at the 5% level. Considering the dropouts, a total of 50 patients (n=25 each group) will be recruited for the study.

Method: - Study subjects will be recruited from the pool of patients enrolling in the Outpatient department meeting the inclusion criteria in the Post Graduate Department of Conservative Dentistry & Endodontics at PGIDS, Rohtak ,Haryana. Study will be performed after obtaining due ethical clearance from Institutional Ethical Committee of PGIDS. Patients are randomly divided into 2Dimensional periapical radiography (PA) group and 3Dimensional Cone beam computed tomography (CBCT) group. Preoperative radiographs (both PA radiography and CBCT) will be taken and periapical surgical procedures will be carried out under operating microscope by the standardized treatment methods.

Surgical Technique:

With the exception of incisions, flap elevation and suturing, all surgical procedures will be performed under operating microscope in an operating room under 8x to 16x magnification.

The full thickness (mucoperiosteal flap) will be reflected under aseptic conditions -

1. Preoperative mouth rinse with 0.2% chlorhexidine mouthwash will be used.
2. Local anaesthesia with lidocaine 2% with epinephrine 1:1,00,000 will be achieved.
3. Buccal intrasulcular incision will be given up to the alveolar crest including one tooth mesial to the lesion & one tooth distal to the lesion, using no.15 BP blade.
4. Mesial and distal vertical releasing incision will be given.
5. Full thickness flap will be gently reflected towards the apical area by periosteal elevator. The flap will be frequently irrigated with sterile saline to prevent dehydration of periosteal surface.
6. After complete elevation of the flap, bone cutting is done using bur and complete debridement of the bony lesion will be performed by surgical curettes For additional hemostasis during surgery cotton pellets soaked in 0.1% epinephrine will be applied topically as required.
7. A 2-3mm root tip with a 0º to 10º bevel angle will be resected with cylindrical surgical carbide bur at high speed with sterile water coolant.
8. Root end preparations extending 3mm into the canal space along the long axis of the root will be made using piezoelectric ultrasonic retrotips in both groups.
9. Isthmuses, fins, and other significant anatomic irregularities will be identified in high magnification and will be treated with the ultrasonic instruments.
10. Root end filling will be done with mineral trioxide aggregrate (MTA). The adaptation of the filling material to the canal apical walls will be confirmed with the aid of an operating microscope at high magnification.
11. Later wound site will be closed and sutured with 4-0 silk suture after irrigating the defect properly.

Post - Operative Follow-Up:

Clinical and 2D periapical radiographic examinations will be performed every 3, 6, 9 and 12 months by assessing the same parameters as baseline except that PD, CAL will not be measured until 12 months .CBCT scan will be done at 12 months follow up . Routine examination procedure will be used to evaluate any evidence of clinical signs and/or symptoms. Postoperative complications and Oral Health Related Quality of Life (OHQoL) questionnaire response will be assessed.

Healing Outcome measurement:

2D Radiographic healing will be assessed by the criteria followed by Rud et al (1972) and Molven et al (1987) Score 1 - Complete healing, defined by re-establishment of the lamina dura Score 2 - Incomplete healing (scar tissue) Score 3 - Uncertain healing Score 4 - Unsatisfactory healing (failure)

Patient assessment of quality of life following surgical endodontic treatment:

Each patient received a questionnaire to fill out for each day starting the day of surgery for 7 days postoperatively. The questionnaire consisted of 15 questions in which patients were to evaluate their quality of life with the 5-point Likert- type scale, ranging from 1 (not at all) to 5 (very much).

3 Dimensionally at 12 months of follow up periapical healing will be assessed by modified PENN 3D criteria: Score 1 - Complete healing Score 2 - Limited healing Score 3 - Uncertain healing Score 4 - Unsatisfactory healing

ELIGIBILITY:
Inclusion Criteria:

* Patient willingness to participate in the study.
* Patient's age more than 18 years.
* Failed root canal treated permanent teeth with post-treatment apical periodontitis requiring treatment.
* Patients referred for periapical surgery of permanent teeth because of separated instrument fragment, overextended root canal filling material or any other idiopathic reasons.
* Radiographic evidence of periapical radiolucency in failed root canal treated teeth.
* American classification of anesthesiologists (ASA) Class I or ASA Class 2 according to ASA classification.

Exclusion Criteria:

* Positive history of antibiotic use within past three months of the treatment.
* Positive history of analgesic use within the past 7 days.
* Procedural errors in previous root canal treatment which are not manageable.
* Patients who are pregnant, diabetic, having human immunodeficiency virus infection or other immune compromising conditions, had serious medical illness or requiring antibiotic premedication.
* Patients with unrestorable lesions, fractures involving the root and periodontium, and/or periodontally compromised teeth.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Postoperative healing | 12 months
  Radiographic healing will be assessed in periapical radiography and CBCT after 12 months

SECONDARY OUTCOMES:
Quality of life assessment | till 1 wek after surgery
  likert scale of 1 to 5 1- not at all 5 - very much

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Science, Rohtak, Haryana, India

REFERENCES:
- [Derived] Gurusamy K, Duhan J, Tewari S, Sangwan P, Gupta A, Mittal S, Kumar V, Arora M. Patient-centric outcome assessment of endodontic microsurgery using periapical radiography versus cone beam computed tomography: A randomized clinical trial. Int Endod J. 2023 Jan;56(1):3-16. doi: 10.1111/iej.13837. Epub 2022 Oct 2. PMID 36135595